CLINICAL TRIAL: NCT00763919
Title: Customized Adherence Enhancement in Bipolar Disorder (CAE in BD)
Brief Title: Customized Medication Adherence Enhancement for Treating Adults With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor of Psychiatry, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R34MH078967-02 (NIH); R34MH078967 (NIH)
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Bipolar Disorder
Keywords: Patient Non-Adherence; Patient Non-Compliance; Patient Nonadherence; Patient Noncompliance; Patient Refusal of Treatment; Refusal of Treatment; Treatment Refusal
MeSH Terms: conditions — Bipolar Disorder; Patient Compliance; Treatment Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Customized Adherence Enhancement (CAE) (Experimental): Participants, all of whom have a history of medication nonadherence, will be assigned to one or more treatment modules based on their individual profiles.
  Treatment Modules:
  Psychoeducation module Substance abuse module Improved communication/rapport with provider module Medication routines management module
  Interventions: Behavioral: Psychoeducation module; Behavioral: Substance abuse module; Behavioral: Improved communication/rapport with provider module; Behavioral: Medication routines management module

INTERVENTIONS:
Behavioral: Psychoeducation module — The psychoeducation module will use psychological and medication education to address opposition to prophylaxis, denial of illness severity or therapeutic effectiveness, negative attitudes toward drugs in general, lack of information about mood stabilizers, and stigma or embarrassment over medications or in relation to the use of complementary or alternative treatments.
Behavioral: Substance abuse module — The substance abuse module will address problematic substance abuse, particularly as it relates to medication adherence.
Behavioral: Improved communication/rapport with provider module — The provider communication and rapport module will improve health care provider communication to address fear of side effects, concern regarding change in appearance, or side effect-related distress.
Behavioral: Medication routines management module — The medication routines management module will develop strategies and behaviors that help create medication adherence routines for those who have difficulties with medication routines or experience outside opposition to medications.

SUMMARY:
In this study, patients with bipolar disorder who do not take their medications as prescribed will receive specialized education and therapy treatment to determine whether the specialized treatment is effective in helping patients to take their medications consistently.

DETAILED DESCRIPTION:
Bipolar disorder (BPD) is a chronic disorder characterized by manic and depressive episodes that disrupt healthy, functional lives. Despite recent advances in medication treatments, many BPD patients do not take their medications. Medication nonadherence is associated with multiple risks, such as relapse, rehospitalization, lengthier hospital stays, and, in some cases, increased risk of suicide. Some studies have shown that treatment adherence in BPD can be improved, particularly through psychological education, development of self-management strategies or behaviors, and ongoing relapse prevention.

This study will examine the effectiveness of medication adherence treatment modules specialized to deal with specific reasons for nonadherence. Participants, all of whom have a history of medication nonadherence, will undergo structured interviews and complete self-report questionnaires to determine individual reasons for nonadherence. Based on their individual profiles, participants will be assigned to one or more of the following intervention modules:

1. Psychoeducation: This module uses education about BPD and related treatment to address patient issues such as opposition to preventive efforts, denial of the need for or effectiveness of medication, negative attitudes toward drugs in general, lack of information about mood stabilizers, and stigma or embarrassment related to BPD treatment.
2. Substance abuse: This module targets substance abuse problems that interfere with medication adherence.
3. Communication with providers: This module addresses fear of medication side effects by improving communication with health care providers.
4. Medication routines management: This module addresses difficulties establishing a medication routine and outside opposition to medications by developing strategies for consistent medication adherence routines.

Each module will involve four 60-minute sessions conducted in a 4- to 6-week period. The study therapist will conduct each of these sessions individually with the participant, combining or coadministering modules in a single session if participants are assigned to more than one module. Depending on which module or modules participants are assigned to, they may also be contacted by phone one to three times by the therapist to complete all module materials.

This study will be conducted in two phases. In the first, an initial group of participants will undergo the module treatments and then participants and therapists will be interviewed about the effectiveness and feasibility of the interventions. This feedback will be used to refine the modules. In the second phase, a second group of participants will undergo treatment in the refined modules and provide more feedback. All participants will continue with their regular treatment while undergoing module treatments.

Participation in this study will last 4 to 6 weeks, with follow-up interviews and assessments ending 6 months after completion of the intervention. In all, there will be five assessments, completed at an initial screening visit, just before treatment, just after treatment, and 3 and 6 months after the completion of treatment. The initial assessments will last 60 to 90 minutes and involve questionnaires and a structured interview. The other four assessments will last 45 to 60 minutes. Treatment adherence, attitudes toward medications, BPD symptoms, and overall functioning will be measured at each assessment. The number of pills used in each participant's prescription bottles will also be counted as a measure of medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bipolar disorder (BPD) Type I or Type II, as determined by a standardized diagnostic interview, the Mini-International Neuropsychiatric Interview (MINI)
* Demonstrated history of poor medication adherence, as determined by self-report or clinician report. In this study, self-reported treatment nonadherence will be identified with the Tablet Routines Questionnaire (TRQ). Poorly adherent individuals will be defined as those who miss 30% or more of medication within either the past week or past month (those missing 30% or more within past week will be considered to be nonadherent over the past month). Clinician-assessed nonadherence will be identified via a clinician version of the TRQ to identify nonadherence of 30% or more over the past 30 days.
* BPD of at least 2 years' duration
* Treatment with medication to stabilize mood for at least 6 months

Exclusion Criteria:

* Unable/unwilling to participate in psychiatric interviews, as based on the clinical opinion of the investigator or the treating clinician
* High risk of suicide, as seen in factors such as active suicidal ideation, recent suicide attempt, or current intent or plan
* Inability to speak English
* Individuals who have participated in Project 1, Personal Adherence Evaluation of Individuals Receiving Treatment for Bipolar Disorder (PAE in BD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- Connections, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Customized Adherence Enhancement (CAE): Participants, all of whom have a history of medication nonadherence, will be assigned to one or more treatment modules of Customized Adherence Enhancement based on their individual profiles.
Period: Overall Study
Arm/Group | Customized Adherence Enhancement (CAE)
Started | 43
Completed | 30
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Change in Treatment Adherence Within the Past Month as Measured by the Tablet Routines Questionnaire
Description: The minimum score is 0 and the maximum score is 100. A higher score implies poorer treatment adherence.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 28
units on a scale | -27.8 (6.5)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 6 months and baseline equals zero; Test type: Superiority or Other; p < .001, Sign test

2. Primary Outcome: Change in Treatment Adherence Within the Past Week as Measured by the Tablet Routines Questionnaire
Description: The minimum score is 0 and the maximum score is 100. A higher score implies poorer treatment adherence.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 28
units on a scale | -20.6 (8.2)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .01, Sign test

3. Primary Outcome: Change in Treatment Adherence as Measured by the Morisky Scale
Description: The minimum score is 0 and the maximum score is 4. A higher score implies poorer treatment adherence.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 28
units on a scale | -1.7 (.29)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 6 months and baseline equals zero; Test type: Superiority or Other; p < .001, Sign test

4. Primary Outcome: Change in Treatment Adherence Within the Past Month as Measured by the Tablet Routines Questionnaire
Description: The minimum score is 0 and the maximum score is 100. A higher score implies poorer treatment adherence.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 33
units on a scale | -28.9 (6.0)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p < .001, Sign test

5. Secondary Outcome: Change in Attitude as Measured by the Attitude Toward Mood Stabilizers Questionnaire (AMSQ)
Description: The AMSQ is a modification of the Lithium Attitudes Questionnaire. The minimum score is 0 and the maximum score is 19. A higher score implies a poorer attitude.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 31
units on a scale | -4.1 (3.2)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p < .001, t-test, 2 sided

6. Secondary Outcome: Change in Attitude as Measured by the Rating of Medication Influences (ROMI)
Description: The minimum score is 0 and the maximum score is 10. A higher score implies a poorer attitude.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | -1.8 (.86)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .042, t-test, 2 sided

7. Secondary Outcome: Change in Depression as Measured by the Hamilton Rating Scale for Depression (HAM-D)
Description: The minimum score is 0 and the maximum score is 52. A higher score implies a worse condition.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | -2.5 (1.4)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .044, Sign test

8. Secondary Outcome: Change in Symptoms of Bipolar Disorder as Measured by the Young Mania Rating Scale (YMRS)
Description: The minimum score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | -4.9 (1.4)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .002, t-test, 2 sided

9. Secondary Outcome: Change in Symptoms of Bipolar Disorder as Measured by the Brief Psychiatric Rating Scale (BPRS)
Description: The minimum score is 18 and the maximum score is 126. A higher score implies a worse condition.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | -8.0 (2.1)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .001, Sign test

10. Secondary Outcome: Change in Global Psychopathology as Measured by the Clinical Global Impression for Bipolar Disorder (CGI-BP)
Description: The minimum score is 1 and the maximum score is 7. A higher score implies a worse condition.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | -.90 (.25)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .001, t-test, 2 sided

11. Secondary Outcome: Change in Functional Status as Measured by the Global Assessment of Functioning (GAF) Scale
Description: The minimum score is 1 and the maximum score is 100. A higher score implies higher functioning.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | 6.7 (1.8)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .001, t-test, 2 sided

12. Secondary Outcome: Change in Perception of Physical Health as Measured by the 12-item Short Form Health Survey (SF-12)
Description: The minimum score is 1 and the maximum score is 99. A higher score implies higher perceived physical health.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 27
units on a scale | .48 (2.2)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .827, t-test, 2 sided

13. Secondary Outcome: Change in Perception of Mental Health as Measured by the 12-item Short Form Health Survey (SF-12)
Description: The minimum score is 1 and the maximum score is 99. A higher score implies higher perceived mental health.
Time Frame: baseline and 6 months
Population: Number of participants for analysis was based on all available data at the six month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 27
units on a scale | 6.9 (2.0)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 6 months and baseline equals zero; Test type: Superiority or Other; p = .002, t-test, 2 sided

14. Secondary Outcome: Change in Depression as Measured by the Hamilton Rating Scale for Depression (HAM-D)
Description: The minimum score is 0 and the maximum score is 52. A higher score implies a worse condition.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 32
units on a scale | -1.4 (1.2)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .246, t-test, 2 sided

15. Secondary Outcome: Change in Symptoms of Bipolar Disorder as Measured by the Young Mania Rating Scale (YMRS)
Description: The minimum score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 32
units on a scale | -2.8 (1.7)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .101, Sign test

16. Secondary Outcome: Change in Symptoms of Bipolar Disorder as Measured by the Brief Psychiatric Rating Scale (BPRS)
Description: The minimum score is 18 and the maximum score is 126. A higher score implies a worse condition.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 32
units on a scale | -6.6 (2.4)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .003, Sign test

17. Secondary Outcome: Change in Global Psychopathology as Measured by the Clinical Global Impression for Bipolar Disorder (CGI-BP)
Description: The minimum score is 1 and the maximum score is 7. A higher score implies a worse condition.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 32
units on a scale | -.47 (.27)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .096, t-test, 2 sided

18. Secondary Outcome: Change in Functional Status as Measured by the Global Assessment of Functioning (GAF) Scale
Description: The minimum score is 1 and the maximum score is 100. A higher score implies higher functioning.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 32
units on a scale | 3.5 (.39)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .072, Sign test

19. Secondary Outcome: Change in Attitude as Measured by the Attitude Toward Mood Stabilizers Questionnaire (AMSQ)
Description: as for outcome 5
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 33
units on a scale | -3.2 (.62)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p < .001, t-test, 1 sided

20. Secondary Outcome: Change in Attitude as Measured by the Rating of Medication Influences (ROMI)
Description: The minimum score is 0 and the maximum score is 10. A higher score implies a poorer attitude.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 33
units on a scale | -1.6 (.88)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .078, t-test, 2 sided

21. Primary Outcome: Change in Treatment Adherence Within the Past Week as Measured by the Tablet Routines Questionnaire
Description: The minimum score is 0 and the maximum score is 100. A higher score implies poorer treatment adherence.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 33
units on a scale | -21.8 (6.8)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .002, Sign test

22. Secondary Outcome: Change in Perception of Physical Health as Measured by the 12-item Short Form Health Survey (SF-12)
Description: The minimum score is 1 and the maximum score is 99. A higher score implies higher perceived physical health.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 32
units on a scale | 1.1 (1.9)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .562, t-test, 2 sided

23. Secondary Outcome: Change in Perception of Mental Health as Measured by the 12-item Short Form Health Survey (SF-12)
Description: The minimum score is 1 and the maximum score is 99. A higher score implies higher perceived physical health.
Time Frame: baseline and 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 32
units on a scale | 3.8 (2.4)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = .12, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years and 3 months
Arm/Group | Customized Adherence Enhancement (CAE)
Serious Adverse Events (participants affected / at risk) | 8/43
Other Adverse Events (participants affected / at risk) | 4/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Customized Adherence Enhancement (CAE) (N=43)
worsening mania (Psychiatric disorders) | 2 (2)
death (Social circumstances) | 1 (1) — As of the last follow-up, the cause of the participant's death was under investigation by authorities.
worsening anxiety/panic attack (Psychiatric disorders) | 1 (1)
suicidal thoughts (Psychiatric disorders) | 2 (2)
incarcerated (Social circumstances) | 1 (1) — The participant was incarcerated for domestic violence.
boils beneath arms (hydronitis) (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Customized Adherence Enhancement (CAE) (N=43)
Suicidal thoughts without plan (Psychiatric disorders) | 1 (1)
mental instability (Psychiatric disorders) | 1 (1)
Worsening depression (Psychiatric disorders) | 1 (1)
Worsening mania (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No